CLINICAL TRIAL: NCT00441818
Title: A Phase I/II, Non-Randomized,Multiple-Dose,Dose Escalation Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of TNX-650 in Patients With Refractory Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of TNX-650 to Treat Refractory Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanox (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-650.101
Record Dates: First submitted 2006-05-17; First posted 2007-03-01 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2007-02

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TNX-650

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of TNX-650 for Injection when administered to patients with refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Hodgkin's lymphoma (HL) is a lymphoid malignancy that accounts for approximately 7,000 to 8,000 new cancer cases per year in the United Sates. It occurs with a bimodal age-incidence distribution peaking in the 15- to 30-year old and 50- to 60-year old age groups. The pathological hallmark of the disease is the presence of malignant Reed Sternberg (RS) cells. Reed-Sternberg cells are interspersed among a heterogeneous population of non-malignant reactive cells, including T cells, eosinophils, neutrophils, B lymphocytes, plasma cells, histiocytes, fibroblasts, and stromal cells.

While more than 80% of patients will respond to initial radiotherapy or combination chemoradiotherapy, some patients will experience early relapse after initial therapy or be refractory to first-line therapy. These patients may be treated with second-line therapy, which may include autologous bone marrow transplantation (BMT). Patients with HL who relapse after first- and second-line therapy, or who are refractory to therapy, with or without autologous BMT, have a poor prognosis. The long-term event-free survival rate in this patient group is less than 10%; median survival is 16 months. At present, these patients have no treatment options other than investigational therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of relapsed or refractory classical HL
* Age >18 years
* Received and failed potentially curative chemotherapeutic regimens (e.g., ABVD, Stanford V, or BEACOPP)
* Relapsed following autologous bone marrow transplantation (BMT), or are ineligible, or refused BMT
* Completed radiotherapy, chemotherapy, and/or treatment with other investigational agents at least 3 weeks prior to study entry
* Completed autologous BMT (if received) at least 3 months prior to study entry; completed allogeneic BMT (if received); at least 6 months prior to study entry
* Eastern Cooperative Oncology Group (ECOG) status of <2
* Life expectancy of >3 months
* Laboratory data:

  * Platelet count >50,000/mm3
  * Hemoglobin >9.0 g/dL (may be maintained by transfusion)
  * Absolute neutrophil count >1000/mm3
  * ALT/AST <2.5 times the upper limit of normal (ULN)
  * Total bilirubin <1.5 times ULN
  * Creatinine <1.5 mg/dL
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening; subjects must agree to use a medically appropriate form of birth control from screening until 6 months after the last dose of study medication
* Ability to provide written informed consent

Exclusion Criteria:

* Any significant diseases (other than HL) or clinically significant findings, including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the subject from participating in the study
* History or clinical evidence of cnetral nervous system (CNS) HL
* Received allogeneic BMT
* Received growth factor support or transfusions to achieve hematology entry criteria (platelets, hemoglobin, absolute neutrophil count)
* Major surgery within 4 weeks prior to study entry
* Known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation
* Known history of another primary malignancy that has not been in remission for at least 5 years. Non-melanoma skin cancer and cervical carcinoma in situ or squamous intraepithelial lesions (e.g., cervical intraepithelial neoplasia [CIN] or prostatic intraepithelial/intraductal neoplasia [PIN]) are allowed.
* Any active viral, bacterial, or systemic fungal infection within 4 weeks prior study entry
* Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV)
* Histry of significant chronic or recurrent infections requiring treatment
* Receiving systemic steroids exceeding 10 mg prednisone or equivalent, or unstable on steroid medication, during the 3 weeks immediately preceding enrollment
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2006-05; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of TNX-650 for Injection when administered to patients with refractory Hodgkin's Lymphoma (HL)
To determine the maximum tolerated dose (MTD) of TNX-650 for Injection
To determine the systemic exposure to TNX-650 for Injection in patients with refractory HL
To determine phosphorylated STAT-6 and IL-13Rα1 levels in tumor samples, and serum IL 13 levels, which may be useful as early prognostic indicators of efficacy in later clinical studies
To determine the preliminary efficacy of TNX-650 for Injection at the maximum tolerated dose (MTD) or pharmacologically active dose, if MTD is not reached, based on tumor assessments using computed tomography (CT) or magnetic resonance imaging (MRI), and

SECONDARY OUTCOMES:
To determine the safety profile of TNX-650 for Injection at the MTD
To determine phosphorylated STAT-6 and IL-13Rα1 levels in tumor samples, and serum IL 13 levels, which may be useful as early prognostic indicators of efficacy in later clinical studies
To determine the preliminary efficacy of TNX-650 for Injection at the MTD, based on tumor assessments using CT or MRI, and FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — M.D. Anderson Cancer Center; Craig Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center - Dept. of Lymphoma and Myeloma, Houston, Texas

REFERENCES:
- See also: Tanox, Inc. website — http://www.gene.com/gene/index.jsp